CLINICAL TRIAL: NCT04378348
Title: Prevention Program to Reduce Injury Disparities Among Latino Day Laborers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Maria E Fernandez-Esquer, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HSC-SPH-12-0818
Record Dates: First submitted 2020-05-04; First posted 2020-05-07 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-05

CONDITIONS: Work-related Injury
Keywords: latino day laborers
MeSH Terms: interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Motivational Interview (Experimental)
  Interventions: Behavioral: Motivational Interview (MI)
- Participatory Group Activity (Experimental)
  Interventions: Behavioral: Participatory Group Activity
- Control Condition (Placebo Comparator)
  Interventions: Behavioral: Control Condition

INTERVENTIONS:
Behavioral: Motivational Interview (MI) — The MI dialogue will begin with an introduction where the LDL is asked about the type of work he does and his concerns regarding dangers in his workplace. This will be followed by a decisional balance exercise where the interviewer will engage the LDL in thinking about the pros and cons of taking jobs with many dangers and jobs with less dangers. Using a figure of a traffic light, the interviewer will proceed to measure how important it is for the LDL to reduce the dangers in his work place and identify his reasons for its importance. Next, the interviewer will measure the LDL's level of confidence in his ability to reduce the dangers in his workplace.Together, they will develop a plan to reduce the dangers in the workplace. Finally, the interviewer will summarize the safety plan to the LDL and will explain that the team will return to the corner in one month to see how the implementation of his plan went and to conduct a post-test survey
  Arms: Motivational Interview
Behavioral: Participatory Group Activity — Participants will view a figure of a pyramid representing the steps they can take to reduce the dangers in their workplace and the things that are in their control to reduce the dangers followed by pictures of dangerous work environments. They will be engaged in hazard identification and situational awareness by identifying and sharing out loud the dangers they see in the picture. Participants will also engage in problem solving by coming up with strategies they could use to reduce the dangers they identified in the picture and will measure their level of confidence in their ability to implement the strategies they have come up with, should they find themselves in a similar work situation. The group facilitator will summarize what the group has said and what they have learned during the group activity and will ask participants to voluntarily make a personal promise to take concrete steps to reduce the dangers at their work.
  Arms: Participatory Group Activity
Behavioral: Control Condition — At control corner sites, we will recruit another 35 Latino day laborer participants.Participants in the control group will receive OSHA pamphlets with standard workplace safety and health information. During our needs assessment survey, we collected information regarding workrelated injuries. Results from this survey indicate the following 4 categories are the highest cause of injury among surveyed Latino day laborers: 1) moving heavy objects, 2) falls, 3) being struck by falling or lying objects, and 4) serious cuts. The OSHA materials that will be distributed to participants will include safety and health information regarding these four topics. Furthermore, given that the LDL are continuously exposed to the sun (e.g., at the corner while waiting for work, at work, and on their way to and from work), heat exposure will also be included in the OSHA materials.
  Arms: Control Condition

SUMMARY:
The purpose of this study is to Identify intervention priorities using a corner-based needs assessment to document occupational and psychosocial risk and protective factors that increase Latino day laborers(LDL) risk for injury and to design a culturally responsive and context appropriate Occupational Safety and Health Administration (OSHA) 10-based safety intervention that also addresses psychosocial risks to reduce LDL injuries and collaboratively pilot a corner-level intervention and conduct an evaluation to assess the safety program's feasibility and acceptability as determined by the extent to which we can recruit, retain and follow-up LDL over the course of the study.

ELIGIBILITY:
Inclusion Criteria:

* Latino
* identified at a "corner" located in the Houston metropolitan area
* currently looking for work at a corner

Exclusion Criteria:

* not of Hispanic/Latino background
* being unable to participate in the survey due to alcohol or drug use impairment.

Min Age: 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2015-10-26 (Actual); Primary Completion 2015-11-03 (Actual); Study Completion 2015-12-08 (Actual)

PRIMARY OUTCOMES:
Exposure to dangers in the workplace as assessed by a questionnaire | Baseline
  The questionnaire asks how often the participant has worked with asbestos, lead paint, Clorox, oil paint, solvents (such as paint thinner), insecticides (such as Raid), glue or adhesive, equipment that creates dust, gasoline or diesel, and cleaning solutions. Each of 10 items on the questionnaire are rated as 1 Never, 2 Sometimes, 3 Many Times, or 4 All the Time, with a total score ranging from 10 to 40, with higher scores indicating greater exposure to dangers in the workplace.
Exposure to dangers in the workplace as assessed by a questionnaire | 1 month
  The questionnaire asks how often the participant has worked with asbestos, lead paint, Clorox, oil paint, solvents (such as paint thinner), insecticides (such as Raid), glue or adhesive, equipment that creates dust, gasoline or diesel, and cleaning solutions. Each of 10 items on the questionnaire are rated as 1 Never, 2 Sometimes, 3 Many Times, or 4 All the Time, with a total score ranging from 10 to 40, with higher scores indicating greater exposure to dangers in the workplace.
Number of participants who had a severe injury or illness in the past month related to their job as a day laborer | Baseline
  Severe injury or illness is defined as an injury or illness where the participant missed work because o the injury or illness, the participant should not have gone to work but you did anyway, or the participant had to receive medical attention from a doctor or a clinic.
Number of participants who had a severe injury or illness in the past month related to their job as a day laborer | 1 month
  Severe injury or illness is defined as an injury or illness where the participant missed work because o the injury or illness, the participant should not have gone to work but you did anyway, or the participant had to receive medical attention from a doctor or a clinic.

SECONDARY OUTCOMES:
Number of participants who had anything happen to them at work in the past month that almost caused them to be injured or made them feel that they could have been injured | Baseline
Number of participants who had anything happen to them at work in the past month that almost caused them to be injured or made them feel that they could have been injured | 1 month
Feasibility and acceptability as indicated by number of participants recruited to the study | Baseline
Feasibility and acceptability as indicated by number of participants retained in the study | 1 month
Feasibility and acceptability as indicated by number of participants who completed the one month follow up | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Maria Fernandez-Esquer, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fernandez-Esquer ME, Atkinson JS, Hernandez RA, Aguerre CF, Brown LD, Reininger B, Ojeda MA, Field C, Rhoton JM, Da Silva CE, Diamond PM. Vales+Tu: a cluster-randomized pilot study to reduce workplace injuries among US Latino day laborers. Health Promot Int. 2022 Dec 1;37(6):daac163. doi: 10.1093/heapro/daac163. PMID 36367426